CLINICAL TRIAL: NCT00505583
Title: A Randomized, Double-Blind, Triple-Dummy, 3-Period Crossover Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of a New Formulation of MOA-728 in Subjects on Stable Methadone Maintenance
Brief Title: Study Evaluating Oral MOA-728 in Subjects on Methadone Therapy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Jeff Cohn, Salix Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3200A3-1110
Record Dates: First submitted 2007-07-16; First posted 2007-07-23 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Methadone-maintenance Subjects

INTERVENTIONS:
Drug: MOA-728

SUMMARY:
To evaluate the effects of single oral doses of MOA-728 compared to a positive control in subjects on methadone therapy.

ELIGIBILITY:
Inclusion:

1. Healthy men or women, aged 18 to 65 years.
2. History of methadone treatment for at least 1 month, at a dose >=30 and <=140 mg/day.

Exclusion:

1. History or active presence of clinically important medical disease.
2. Allergy to opioids.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-07; Primary Completion 2007-12 (Estimated); Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
To characterize the pharmacodynamics of single oral doses of MOA-728 compared to a positive control of MOA-728 administered intravenously in subjects on stable methadone maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Cohn, Study Director — Bausch Health Americas, Inc.
Locations (1):
- Gainesville, Florida, United States